CLINICAL TRIAL: NCT02758223
Title: Prophylactic Application of Donor-derived Central Memory T Lymphocytes (TCM) After Allogeneic HSCT to Prevent Infectious Complications
Brief Title: Prophylactic Application of Donor-derived TCM After Allogeneic HSCT
Acronym: PACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACT2014-001; 2015-001522-41 (EudraCT Number)
Record Dates: First submitted 2016-02-25; First posted 2016-05-02 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cryopreservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Experimental: TCM allogeneic humane central memory T cells, cryopreserved Solution for injection (intravenous use) up to 65*10^4 TCM /kg body weight patient will receive investigational product 3 times (Day 30, Day 60, Day 90 after alloHSCT)
  Interventions: Biological: TCM allogeneic humane central memory T cells, cryopreserved

INTERVENTIONS:
Biological: TCM allogeneic humane central memory T cells, cryopreserved — Experimental: TCM allogeneic humane central memory T cells, cryopreserved Solution for injection (intravenous use) up to 65*10^4 TCM /kg body weight patient will receive investigational product 3 times (Day 30, Day 60, Day 90 after alloHSCT)

SUMMARY:
PACT is a non-randomized multicentre phase I/II study to evaluate the feasibility and safety of the prophylactic administration of donor derived TCM. Patients with Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) who are planned to undergo a HLA -matched (9/10 or 10/10) allogeneic hematopoietic stem cell transplantation and who are either 50+ years old or have a high comorbidity score are included according to criteria as described below. TCM will be applied in escalating doses to a maximum of 30 patients who have received T cell depleted Human leukocyte antigen (HLA)-matched alloHSCT grafts and qualify for TCM transfer.

DETAILED DESCRIPTION:
One of the major challenges in the field of allo-SCT is to find a balance between the harmful induction of graft-versus-host disease (GVHD) and the beneficial graft-versus-leukemia (GVL) response, both mediated by donor T cells recognizing antigens expressed on cells of the recipient. Complete removal of T cells from the graft results in abrogation of severe GVHD, but is also frequently associated with removal of the immunity against infectious agents and the anti-tumor efficacy (GVT effect), which is reflected by an increased incidence of infectious complications and (early) disease relapses after T cell depleted allo-SCT. The investigators hypothesize that the prophylactic adoptive transfer of donor-derived central memory T cells is a safe and tolerable method to improve overall survival after HSCT.

TCM are administered in escalating doses at day 30, day 60 and day 90 posttransplant to prevent infectious complications and early relapse or disease progression.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Male or female patients with Hematopoietic Cell Transplant-Co-morbidity Index (HCT-CI) score (Sorror) ≥3 AND/or Age 50 years or older
* Primary or secondary AML Month 0, Month 1, Month 2, Month 4, Month 5, Month 6 and Month 7, in Complete Remission (CR) (<5% blasts in bone marrow (BM)) irrespective of the cytogenetic or molecular risk profile or MDS up to Refractory anemia with excess of blasts 2 (RAEB-2) (maximal 20% blasts in bone marrow)
* Planned alloHSCT with Cluster of Differentiation 34+ (CD34+)-purified stem cell grafts after conditioning with fludarabine-melphalan-thio-thepa-ATG (ATG=Antithymocyte globulin)
* HLA-matched stem cell donor (9-10/10, maximal 1 allel- or antigen mismatch allowed) without aberrant CD45RA (=Cluster of Differentiation) expression

Additional patient inclusion criteria: Treatment phase patients at day 30 +/-5 after alloHSCT:

-Stable engraftment of the allogeneic graft (granulocytes > 0.5*109/L)

Donor

* Donor must have met requirements of European Union (EU) Tissue and Cells Directive (2004/23/EC) (see below)
* Healthy donor - having passed medical examination for stem cell donation
* Donor must fulfill the requirements for allogeneic donor blood testing according to Richtlinie zur Herstellung und Anwendung von hämatopoetischen Stammzellzubereitungen (SC-Richtlinie (RILI) der Bundesärztekammer; 08/2014)
* Donor informed consent for the additional non-mobilized apheresis
* Written informed consent of the patient

Exclusion Criteria:

* Patient
* Disease-specific treatment foreseen in the first 6 months after alloHSCT
* Patients with AML M3
* Pregnant or lactating women
* Severe psychological disturbances
* Positive serology for Human immunodeficiency virus (HIV), Syphilis, West Nile Virus (WNV)
* Participation in another interventional clinical trial during or within 4 weeks before study entry Additional patient exclusion criteria: Treatment phase patients at day 30 +/-5 after alloHSCT:
* Disease specific treatment foreseen in the first 6 months after alloHSCT
* Acute GVHD > grade I for which immune suppressive treatment is given
* Progressive disease for which therapy is needed
* Use of > 0,5 mg/kg bw prednisone a day
* Life expectation < 12 weeks
* End stage irreversible multi-system organ failure

Donor

* Donor pregnant or lactating
* Donors with aberrant CD45RA isoform expression
* General exclusion criteria for stem cell donation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of acute GVHD > overall grade II or death | during three months after the infusion of the T cell product
  Toxicity of the infusion will be evaluated by the cumulative incidence of acute GVHD > overall grade II or death during three months after the infusion of the T cell product.

SECONDARY OUTCOMES:
Appearance or Expansion of antigen specific T cells measured in specific T cells per mikroliter | during 9 months after first infusion
  the determination of appearance or expansion of antigen specific T cells (measured in specific T cells per mikroliter) from donor derived TCM during 36 weeks (9 months) after the first infusion of study medication.
Clinical signs of viral infections - fever in °celsius | During 10 months after first application until study end (per patient)
  Clinical signs of viral infections - fever in °celsius
Incidence of relapse | During 10 months after first application until study end (per patient)
Incidence of bacterial and fungal infections | During 10 months after first application until study end (per patient)
Incidence of GvHD grade II-IV | During 10 months after first application until study end (per patient)
Donor chimerism in bone marrow and peripheral blood measured in % of nucleated cells | During 10 months after first application until study end (per patient)
Incidence of viremia and clinical manifestations of virus-related organ manifestations (Cytomegalovirus (CMV), Eppstein-Barr virus (EBV), Adenovirus, Herpes Simplex Virus (HSV), Varicella-Zoster Virus (VZV)) | During 10 months after first application until study end (per patient)
quantification of CMV specific T cells by multimer staining and ics (copies / ml) | before transfer of the first TCM dose (Month 0) and at Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8 and Month 9 after first TCM transfer.
  Efficacy of the transfer of TCM will be evaluated by quantification of CMV specific T cells by multimer staining and ics before transfer of the first TCM dose (Month 0) and at Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8 and Month 9 after first TCM transfer.
quantification of EBV specific T cells by multimer staining and ics (copies / ml) | before transfer of the first TCM dose (Month 0) and at Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8 and Month 9 after first TCM transfer.
  Efficacy of the transfer of TCM will be evaluated by quantification of EBV specific T cells by multimer staining and ics before transfer of the first TCM dose (Month 0) and at Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8 and Month 9 after first TCM transfer.
quantification of Adenovirus specific T cells by multimer staining and ics (copies / ml) | before transfer of the first TCM dose (Month 0) and at Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8 and Month 9 after first TCM transfer.
  Efficacy of the transfer of TCM will be evaluated by quantification of Adenovirus specific T cells by multimer staining and ics before transfer of the first TCM dose (Month 0) and at Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8 and Month 9 after first TCM transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Götz U Grigoleit, PhD, Principal Investigator — University Hospital Wuerzburg- Departement of Medicine II
Locations (1):
- University Hospital Wuerzburg - Department of Medicine II, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No